CLINICAL TRIAL: NCT04975633
Title: USC and Bodyport Remote Heart Failure Management Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael William Fong, Associate Professor of Clinical Medicine, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: HS-21-00032
Record Dates: First submitted 2021-05-24; First posted 2021-07-23 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- BodyPort Cardiac Scale (Experimental): Patient will receive the Bodyport scale with access to Bodyport care services, such as remote monitoring, educational materials, different biomarkers detected by the scale, and online access to their data
  Interventions: Device: Bodyport Cardiac Scale
- Control (No Intervention): Patients will receive usual care and a Bodyport scale that only displays weight and weight change. No other access to care services, features, or materials will be provided during this 90 day period

INTERVENTIONS:
Device: Bodyport Cardiac Scale — Patients will be instructed to take daily measurements for 90 days. Data will be transmitted to Bodyport and concerning findings (weight gain, change of impedance, elevated heart rate) will be reported back to the medical team. The medical team will either choose to act on the information given or continue to observe trends. Interventions may include titration of therapy, change in therapy, fluid restriction, sodium restriction and lifestyle modification
  Arms: BodyPort Cardiac Scale

SUMMARY:
A feasibility study investigating the Bodyport virtual cardiac clinic vs usual care for outpatient heart failure management at Keck Medical Center of USC

DETAILED DESCRIPTION:
Heart failure is a debilitating disease associated with high hospitalization rates which could potentially be curbed by remote patient monitoring. Remote monitoring may allow for the early detection of signs and symptoms of cardiac decompensation, enabling prompt interventions to reduce hospital admission rates or the duration of inpatient stay, and the quality of life of those suffering from heart failure. Recent studies have demonstrated that structured remote patient management interventions can reduce the percentage of days lost to unplanned cardiovascular admissions. The investigators propose assessing the feasibility of a structured virtual cardiac care service leveraging the Bodyport platform to optimize outpatient management of heart failure.

This study will leverage the Bodyport virtual cardiac clinic platform to deliver care for the heart failure patient population at Keck Medical Center of USC. Patients randomized to the intervention arm will receive the Bodyport Cardiac Scale for home monitoring as well as heart failure education and non-clinical support from Bodyport coaches. Daily measurement uploads from the patients will be analyzed and changes in measurement data will be used to guide follow-up and care management, such as diuretic dose adjustments. For this initial feasibility study, the investigators will be focusing on patient and provider satisfaction of the virtual cardiac clinic along with the operational ease of executing this form of care compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HFrEF or HFpEF and hospital discharge for a heart failure exacerbation within 14 days of enrollment.
* 18 years of age or older
* English speaking
* Able to safely stand on the Bodyport scale
* Patients must have a reliable and working phone for communication with the care team
* All patients should have access to the internet via a computer or mobile device to access the Bodyport care platform
* Patients must have a safe and secure place to store the Bodyport device

Exclusion Criteria:

* Weight >375 lbs.
* History of repeatedly missing follow-up appointments or being unreachable by phone
* Inability to stand on the Bodyport scale for the duration needed to capture data
* Patient in jail or currently homeless
* Known or documented noncompliance with medical therapy
* Unable to speak English
* Unable or unwilling to answer survey questions
* History of heart transplantation
* Chronic kidney disease stage IV or V and/or on hemodialysis
* Presence of a ventricular assist device
* Presence of a CardioMEMs pulmonary artery sensor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2024-09-05 (Actual); Study Completion 2024-09-05 (Actual)

PRIMARY OUTCOMES:
Change in quality of life | Up to 14 days after enrollment and approximately 90-days post-enrollment
  Evaluating Kansas City Cardiomyopathy Questionnaire (KCCQ) measurements at the time of hospital discharge and 90-days post-discharge
Scale Adherence | Through study completion, approximately 90 days
  Measure of daily scale adherence

SECONDARY OUTCOMES:
Patient and provider satisfaction | Through study completion, approximately 90 days for patients and an average of 9 months for providers.
  Assessing patient and provider satisfaction with the Bodyport virtual cardiac clinic at USC Keck Medicine through semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Michael W Fong, MD, Principal Investigator — Keck Medical Center of USC
Locations (1):
- Keck Medical Center of USC, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No